CLINICAL TRIAL: NCT04799795
Title: Objective EEG Bed Side Assessment of Impaired Conscious Awareness in Epilepsy
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Gesine Hermann, MD, Scientist in Neuroimaging, University Hospital Schleswig-Holstein
Other Study IDs: D 558/17
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy, Absence
Keywords: interictal activity; impaired consciousness; absence epilepsy
MeSH Terms: conditions — Epilepsy, Absence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy subjects: Age-matched healthy participants will be recruited via flyers at public education facilities and online advertisement. Participants need to be healthy and without central nervous system disorders and substance abuse. The investigators will also exclude pregnant women from the experiment.
- patients with absence epilepsy: Apart from the diagnosis of epilepsy, patients need to be of good health and without central nervous system disorders and substance abuse. The investigators will also exclude pregnant women from the experiment.

SUMMARY:
In this project EEG recordings between healthy participants and those with a diagnosed Absence-epilepsy will be compared. The investigators suggest differences in EEG microstate analysis and neuropsychological parameters related to interictal cognitive impairment in these patients. This projects goal is to derive an EEG-based measure of conscious awareness.

DETAILED DESCRIPTION:
This projects goal is to derive an EEG-based measure of conscious awareness to be applied in the care for epilepsy patients. The established terminology of "ictal" versus "interictal" is deceptive because it suggests that during the "interictal" phase epileptic activity is absent and detrimental mechanisms of the disease are only active during seizures. But evidence exists that cognitive impairment extends to states traditionally considered interictal. The development of an objective, ideally ambulatory test assessing cognitive impairment would not only provide a deeper understanding of the pathology but induce a change in clinical practice: if cognitive impairment could be demonstrated "interictally", this fact would help to weigh treatment effects against potential side-effects.

In this project the investigators will set out to

1. identify EEG markers in healthy volunteers, which reflect the changes in spatial and temporal dynamics of neuronal activity during states of reduced conscious awareness using sleep as an example of a state of reduced conscious awareness;
2. assess with neuropsychological testing reductions in interictal conscious awareness in patients with epilepsy;
3. test, whether markers established under (1) are valid in individuals with epilepsy and interictally reduced conscious awareness (see (2)).

ELIGIBILITY:
Inclusion Criteria:

* age minimum 18 years
* diagnosis of (absence) epilepsy // healthy age-matched controls
* being of good health (besides epilepsy in the case group)

Exclusion Criteria:

* central nervous system disorders (besides epilepsy in the case group)
* substance abuse
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed absence epilepsy at least 18 years old; age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-05-24 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
temporal integration changes according to different sleep states | 3 years
  The investigators develop an EEG-based measure of impaired conscious awareness based on wakefulness and deepening sleep stages which will serve as a model for increasingly impaired conscious awareness. By performing a microstate analysis on EEG data, the investigators hypothesize a decrease of the temporal integration, a prerequisite for conscious awareness, of the EEG gradually from wakefulness to deep sleep.
temporal integration changes in interictal EEG | 3 years
  The investigators apply the aforementioned analysis (leading to Outcome 1) on interictal EEG recordings obtained from patients with diagnosed absence epilepsy. The investigators hypothesize a reduced temporal integration in epilepsies with reduced consciousness.
graph modularity changes according to different sleep states | 3 years
  The investigators will calculate the EEG-based functional connectivity and graph modularity for each sleep state. The investigators hypothesize that during wakefulness, graph modularity will be lower than during the descent to sleep.
graph modularity changes in interictal EEG | 3 years
  The investigators will calculate the EEG-based functional connectivity and graph modularity for the absence epilepsy condition. The investigators hypothesize that impaired consciousness will be reflected in lower graph modularity compared to healthy subjects.

SECONDARY OUTCOMES:
EEG based measures (Outcome 4) correlate with | 3 years
  The investigators hypothesize that the graph modularity level correlates with neuropsychological test scores in the surveyed data of epilepsy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Inken Toedt, Dr. phil. Dipl.-Psych., Principal Investigator — University Hospital Schleswig-Holstein, Kiel; Helmut Laufs, PD Dr. med., Study Director — University Hospital Schleswig-Holstein, Kiel
Locations (1):
- Department of Neurology, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Analysis protocols and analysis scripts will be shared between this studies collaborators through a public platform, probably GitHub. The corresponding repositories will be openly accessible.
  Calculated data will be accessible in the context of planned publications afterwards.
  The collected raw data, therefore IPD won't be shared before the final investigation by the study group.

REFERENCES:
- [Background] Brodbeck V, Kuhn A, von Wegner F, Morzelewski A, Tagliazucchi E, Borisov S, Michel CM, Laufs H. EEG microstates of wakefulness and NREM sleep. Neuroimage. 2012 Sep;62(3):2129-39. doi: 10.1016/j.neuroimage.2012.05.060. Epub 2012 May 30. PMID 22658975
- [Background] Haimovici A, Tagliazucchi E, Balenzuela P, Laufs H. On wakefulness fluctuations as a source of BOLD functional connectivity dynamics. Sci Rep. 2017 Jul 19;7(1):5908. doi: 10.1038/s41598-017-06389-4. PMID 28724928
- [Background] Kuhn A, Brodbeck V, Tagliazucchi E, Morzelewski A, von Wegner F, Laufs H. Narcoleptic Patients Show Fragmented EEG-Microstructure During Early NREM Sleep. Brain Topogr. 2015 Jul;28(4):619-35. doi: 10.1007/s10548-014-0387-1. Epub 2014 Aug 29. PMID 25168255
- [Background] Laufs H, Rodionov R, Thornton R, Duncan JS, Lemieux L, Tagliazucchi E. Altered FMRI connectivity dynamics in temporal lobe epilepsy might explain seizure semiology. Front Neurol. 2014 Sep 11;5:175. doi: 10.3389/fneur.2014.00175. eCollection 2014. PMID 25309503
- [Background] Tagliazucchi E, Crossley N, Bullmore ET, Laufs H. Deep sleep divides the cortex into opposite modes of anatomical-functional coupling. Brain Struct Funct. 2016 Nov;221(8):4221-4234. doi: 10.1007/s00429-015-1162-0. Epub 2015 Dec 9. PMID 26650048
- [Background] Tagliazucchi E, Laufs H. Decoding wakefulness levels from typical fMRI resting-state data reveals reliable drifts between wakefulness and sleep. Neuron. 2014 May 7;82(3):695-708. doi: 10.1016/j.neuron.2014.03.020. PMID 24811386
- [Background] Tagliazucchi E, Roseman L, Kaelen M, Orban C, Muthukumaraswamy SD, Murphy K, Laufs H, Leech R, McGonigle J, Crossley N, Bullmore E, Williams T, Bolstridge M, Feilding A, Nutt DJ, Carhart-Harris R. Increased Global Functional Connectivity Correlates with LSD-Induced Ego Dissolution. Curr Biol. 2016 Apr 25;26(8):1043-50. doi: 10.1016/j.cub.2016.02.010. Epub 2016 Apr 13. PMID 27085214
- [Background] Tagliazucchi E, von Wegner F, Morzelewski A, Brodbeck V, Borisov S, Jahnke K, Laufs H. Large-scale brain functional modularity is reflected in slow electroencephalographic rhythms across the human non-rapid eye movement sleep cycle. Neuroimage. 2013 Apr 15;70:327-39. doi: 10.1016/j.neuroimage.2012.12.073. Epub 2013 Jan 9. PMID 23313420
- [Background] Tagliazucchi E, von Wegner F, Morzelewski A, Brodbeck V, Jahnke K, Laufs H. Breakdown of long-range temporal dependence in default mode and attention networks during deep sleep. Proc Natl Acad Sci U S A. 2013 Sep 17;110(38):15419-24. doi: 10.1073/pnas.1312848110. Epub 2013 Sep 3. PMID 24003146
- [Background] von Wegner F, Tagliazucchi E, Laufs H. Information-theoretical analysis of resting state EEG microstate sequences - non-Markovianity, non-stationarity and periodicities. Neuroimage. 2017 Sep;158:99-111. doi: 10.1016/j.neuroimage.2017.06.062. Epub 2017 Jun 30. PMID 28673879

DOCUMENTS (2):
  • Study Protocol (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT04799795/Prot_000.pdf
  • Informed Consent Form (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT04799795/ICF_001.pdf